CLINICAL TRIAL: NCT00601094
Title: A Phase I Trial of CCL21 Gene Modified Dendritic Cells In Non-Small Cell Lung Cancer
Brief Title: Vaccine Therapy in Treating Patients With Stage IIIB, Stage IV, or Recurrent Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-06-008; UCLA-NCI-7888; 10-000039 (Other: Jonsson CCC)
Record Dates: First submitted 2008-01-10; First posted 2008-01-25 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2017-10

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- experimental arm (Experimental)
  Interventions: Biological: autologous dendritic cell-adenovirus CCL21 vaccine

INTERVENTIONS:
Biological: autologous dendritic cell-adenovirus CCL21 vaccine — Eligible patients will be assigned to a cohort and will receive intratumoral injections of Ad-CCL21-DC in conjunction with tumor sampling.

SUMMARY:
RATIONALE: Vaccines made from a gene-modified virus may help the body build an effective immune response to kill tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of vaccine therapy in treating patients with stage IIIB, stage IV, or recurrent non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the safety, toxicity, and maximum tolerated dose (MTD) of autologous dendritic cell-adenovirus CCL21 vaccine administered as an intratumoral injection in treating patients with stage IIIB, IV, or recurrent non-small cell lung cancer.

Secondary

* To determine the biologic and clinical responses to therapy.
* To determine treatment-related toxicity using the NCI Common Toxicity Criteria.
* To identify the MTD.
* To monitor patients for evidence of autologous dendritic cell-adenovirus CCL21 vaccine-induced cytokines and antigen-specific immune responses.
* To detect immune responses to tumor-associated antigens and vector.
* To assess patients for objective signs of tumor regression (RECIST Criteria).

OUTLINE: This is a dose-escalation study of autologous dendritic cell-adenovirus CCL21 vaccine.

Patients undergo leukapheresis to obtain leukocytes for generation of autologous dendritic cells (DC). Adenovirus carrying the CCL21 gene is added to the dendritic cells to make the vaccine. Approximately 2 weeks after leukapheresis, patients receive an intratumoral injection of autologous dendritic cell-adenovirus CCL21 vaccine under CT-guidance or by bronchoscopy on days 0 and 7. Patients demonstrating a clinical response are eligible to receive a second round of gene transfer at their discretion and in consultation with the FDA.

Cohorts of 3 patients receive escalating doses of autologous dendritic cell-adenovirus CCL21 vaccine until the maximum tolerated dose (MTD) is determined. An additional 12 patients are treated at the MTD.

Patients undergo blood sample collection at baseline and then on days 0, 7, 14, 28, and 56 for safety and immunological studies. Blood samples are analyzed for mycoplasma by PCR; dendritic cell phenotype by flow cytometry; detection of adenovirus CCL21 by nested PCR; and adenoviral antibodies by ELISA. Patients also undergo tissue aspirate or biopsy on days 0 and 7 (during bronchoscopy or CT-guided procedure). Tissue samples are analyzed for immune-modulating cytokines (i.e., IFNγ, CXCL9, and CXCL10) by quantitative RT-PCR; detection of tumor infiltrating leukocytes by immunohistochemistry; CD83+ DC, CXCR3, CCR7, CCL21 and CD3+ T-cells, CD4, and CD8 by flow cytometry; determination of tumor expression of tumor-associated antigen by RT-PCR; and evaluation of immune modulation by ELISPOT assays.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
Inclusion Criteria:

* Adults over the age of 21 capable of giving informed consent
* Pathologically confirmed non-small cell lung cancer (NSCLC)
* Stage IIIB, IV, or recurrent disease
* Progressive disease despite one or more prior chemotherapy regimens as standard of care OR patient refuses standard chemotherapy
* Measurable metastatic disease by RECIST guidelines
* Patients with a major endobronchial lesion in the segmental, lobar, or mainstem bronchus with complete obstruction of the airway may be eligible for bronchoscopic injection provided there is no evidence of respiratory failure (defined as SaO_2 > 90% on room air, PCO_2 < 45 mm Hg, or FEV_1 > 1.0 L)
* Patients with an endobronchial lesion in the segmental bronchus with variable stenosis (not completely obstructed) and not amenable to standard palliative airway treatments (i.e., laser and stenting) may be eligible for bronchoscopic injection if there is no evidence of respiratory failure (defined as SaO_2 > 90% on room air, PCO_2 < 45 mm Hg, or FEV_1 > 1.0 liters)
* Patients with bullous disease may undergo CT-guided transthoracic injection provided the targeted tumor has an intended needle path without crossing bullae
* ECOG performance status 0-2
* BUN ≤ 40 OR serum creatinine ≤ 2
* Serum total bilirubin ≤ 1.5 OR serum transaminases ≤ 2.5 times upper limit of normal (ULN)
* Negative pregnancy test
* Fertile patients must use effective contraception
* More than 14 days since prior acute therapy for viral, bacterial, or fungal infections
* More than 30 days since prior and no concurrent corticosteroids
* More than 30 days since prior radiotherapy, chemotherapy, or noncytotoxic investigational agents

Exclusion Criteria:

* active CNS metastasis (i.e., progression of CNS disease during the past 30 days without intervention)
* evidence of coagulopathy, defined as PT and/or PTT ≤ 1.5 times ULN OR platelets ≥ 100,000/mm^3
* evidence of leukoplakia, defined as absolute neutrophil count ≥ 1,500/mm^3
* evidence of respiratory failure (defined as SaO_2 > 90% on room air, PCO_2 < 45 mm Hg, or FEV_1 > 1.0 L)
* NYHA class III-IV cardiac disease within the past year
* myocardial infarction within the past year
* comorbid disease or medical condition that would impair the ability of the patient to receive or comply with the study protocol
* acute viral, bacterial, or fungal infection that requires specific therapy
* HIV positivity
* hypersensitivity to any reagents used in the study
* signs or symptoms of acute adenoviral infection (i.e., conjunctivitis or documented adenoviral upper respiratory infection)
* prior or concurrent evidence of autoimmune disease
* pregnant or nursing
* prior organ allograft

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-02-26 (Actual); Primary Completion 2017-05-23 (Actual); Study Completion 2017-05-23 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 28 days
Toxicity as measured by NCI Common Toxicity Criteria | 28 days

SECONDARY OUTCOMES:
Disease status at days 28 and 56 | 56 days
Immune response assessment by antigen-specific IFNγ ELISPOT assays on days 0, 28, and 56 | 56 days

CONTACTS AND LOCATIONS:
Overall Officials: Jay M. Lee, MD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (2):
- United States (2):
  - VA Greater Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California